CLINICAL TRIAL: NCT02496325
Title: Ultrasound-guided Pudendal Nerve Block in Children: A Descriptive Study of Feasibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 9397; 2014-A00499-38 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2015-06-23; First posted 2015-07-14 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-06

CONDITIONS: Pudendal Nerve Block
Keywords: Pudendal nerve block; Ultrasound guided; Transperineal puncture; Perineal surgery; children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- perineal technic (Other)
  Interventions: Procedure: Ultrasound guided transperineal pudendal nerve block

INTERVENTIONS:
Procedure: Ultrasound guided transperineal pudendal nerve block — Children under general anesthesia were positioned supine, flexed legs and balls of the feet joined. A 12 MegaHertz (MHz) (38 mm) ultrasound probe was positioned on a horizontal axis passing through the ischial tuberosity, previously palpated.The probe was then moved medially on the axis, until the rectum appeared. Pudendal artery was identified if possible, using colour Doppler. The needle (22 Ga, 50 mm) was then introduced at the middle of the superior edge of the probe, in an out-of-plane approach. Tip of the needle was identified by direct vision, through displacement of adjacent anatomical structures or with saline injection. Nerve stimulation was started after placement of the tip of needle in the ischiorectal fossa, before local anaesthetic injection. After a negative aspiration test, a mix of Ropivacaine 2 % and clonidine 0.2µg/kg was injected in the ischiorectal fossa under ultrasound guidance.

SUMMARY:
Objective: Description of a new transperineal technique of pudendal nerve block (PNB), under ultrasound-guidance.

Methods : Successive inclusions after parental consent of 60 children undergoing perineal surgery under general anesthesia and pudendal nerve block. Data were collected from induction of anesthesia to second post-operative day (24 hrs. after admission in recovery room). Ease of PNB achievement was the primary objective evaluated. Efficiency in preoperative and postoperative period was also reported.

DETAILED DESCRIPTION:
After obtaining parental consent, children aged 1-15 years, physical status score I-III, requiring general anesthesia associated with bilateral pudendal nerve block (PNB) for elective perineal surgery in the investigators' paediatric surgery unit, were successively included. Exclusion criteria were any contraindication to general or loco regional anesthesia, and physical status score IV-V. Management of general anesthesia was standardized. Propofol and/or sevoflurane were used for induction, in association with a continuous infusion of remifentanil at 1µg/kg/min during two minutes. After this delay, airway control was assured through insertion of a tracheal tube or a laryngeal mask. Maintenance of anesthesia was then achieved with Sevoflurane (1.2 MAC) in a mix 02/N2 and remifentanil 0.05 µg/kg/min. Mechanical ventilation parameters were adapted to obtain a normal End-tidal carbon dioxide (EtCO2) (28-34 mmHg). Baseline values of blood pressure and heart rate under general anesthesia without nociceptive stimulation were measured.Ultrasound guided pudendal nerve block was then performed. For each block, data about sonographic identification of anatomical structures, visualization of needle and local anaesthetic spread were collected. The response to nerve stimulation, puncture complications and duration of the procedure were also noted. During perineal operative time, a rise up in blood pressure or in heart rate more than 20% compared to baseline values was considered as a PNB failure. Analgesia was then provided by an incremental increase of remifentanil, to obtain a return to baseline hemodynamic parameters. The maximum rate of infusion of remifentanil was collected. All patients received intravenous post-operative analgesia by acetaminophen 15 mg/kg and ketoprofen 1mg/kg. Rescue analgesia by IV nalbuphine 0.2 mg/kg was administered in recovery room if necessary. Post-operative analgesia by oral acetaminophen associated with ibuprofen, and rescue analgesia with oral tramadol were prescribed. Data on post-operative analgesia were collected up to 24h after recovery room admission.

ELIGIBILITY:
Inclusion Criteria:

1. Patient hospitalized in pediatric surgery unit for elective perineal surgery to which the use of pudendal block is relevant and current practice.
2. patient physical status score I-III classification
3. Patient of both sexes
4. Patient aged 1 year to 15 years of age
5. Patient whose parents have given their informed consent.
6. Patient affiliated to a social security scheme or of such a regime

Exclusion Criteria:

1. Patient who participated in the previous month to a therapeutic trial or currently included in another test
2. Patient with bleeding disorders
3. Patient with infection (Fasciocutaneous subcutaneous) at the puncture area
4. Patient with allergies to local anesthetics
5. patients with a contraindication to general anesthesia

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 196 (Actual)
Dates: Start 2014-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Quality of visualization (with specific scale: good, medium, bad quality) of local anesthetic injection within the ischiorectale pit under ultrasound. | intraoperative

SECONDARY OUTCOMES:
Quality of visualization (with specific scale: good, medium, bad quality) of target anatomical structures, of needle tip | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle IG GAUDET-FERRAND, MD, Principal Investigator — Department of Anesthesia Resuscitation at the Hospital Lapeyronie in Montpellier
Locations (1):
- University hospital Lapeyronie, Montpellier, France